CLINICAL TRIAL: NCT04283149
Title: A Multicenter Clinical Evaluation of the EVO/EVO+ Visian® Implantable Collamer® Lens
Brief Title: Multicenter Clinical Trial of a Phakic Implantable Collamer® Lens (ICL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Staar Surgical Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP19-01
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Myopia; Myopic Astigmatism
Keywords: Nearsightedness; Phakic intraocular lens (IOL); ICL; Toric ICL; EVO; EVO+; Visian
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: All enrolled eyes will undergo phakic eye surgery to have one of the available implantable collamer lenses EVO or EVO+ (spherical or toric) ICL implanted in their primary eye. Fellow eye surgery will occur between 7 and 14 days after primary eye surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Primary Eyes (Experimental): First implanted eyes of enrolled participants
  Interventions: Device: EVO/EVO+ Visian ICL
- Fellow Eyes (Experimental): Second implanted eyes of enrolled participants
  Interventions: Device: EVO/EVO+ Visian ICL

INTERVENTIONS:
Device: EVO/EVO+ Visian ICL — The investigational lenses are intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens.

SUMMARY:
This objective of this study is to evaluate the safety, and to collect supportive data on effectiveness of the EVO/EVO+ Visian® Implantable Collamer® Lens (ICL) in study participants who have a diagnosis of myopia or myopia with astigmatism. Primary study analysis will be evaluated when 300 primary eyes complete 6 months of follow-up. Final study analysis will be assessed when all treated eyes complete 36 months of follow-up.

DETAILED DESCRIPTION:
This study will be conducted at up to 20 clinical sites in the United States by surgeons qualified by training and experience to implant STAAR ICLs.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to high myopia or myopic astigmatism correctable with available EVO/EVO+ ICL powers.
* Stable refractive history within 0.50 D each cylinder and spherical equivalent (SE) for 1 year prior to implantation.
* Able and willing to return for scheduled follow-up examinations after surgery.
* Able to read, understand and provide written informed consent on the Institutional Review Board (IRB)-approved informed consent form (ICF) and provide authorization as appropriate for local privacy regulations.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Insulin-dependent diabetes or diabetic retinopathy.
* History of previous ocular surgery.
* Cataract of any grade.
* Monocular.
* Pregnant or nursing women, or those who plan to become pregnant over the course of this clinical study.
* Other protocol-specified exclusion criteria may apply.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 327 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Egamino, PhD, Study Director — VP, Global Clinical Affairs
Locations (14):
- United States (14):
  - Barnett Dulaney Perkins, Phoenix, Arizona
  - Aloha Laser Vision, LLC, Honolulu, Hawaii
  - Price Vision Group,, Indianapolis, Indiana
  - Durrie Vision, Overland Park, Kansas
  - Solomon Eye Physicians and Surgeons/Bowie Vision Institute, Bowie, Maryland
  - Brinton Vision, St Louis, Missouri
  - Kugler Vision, PC, Omaha, Nebraska
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Kremer Eye Center, King of Prussia, Pennsylvania
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Key-Whitman Eye Center, Dallas, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - Hoopes Vision/Hoopes, Durrie, Rivera Research, Draper, Utah
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 327 subjects were enrolled and treated at 14 clinical sites in the US. The first enrolled subject underwent surgery in the primary eye in January 2020 and the last eye was implanted in December 2020.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Primary Eyes | Fellow Eyes
Started | 327; 327 eyes | 327; 302 eyes
Postoperative Month 6 | 321; 321 eyes | 321; 298 eyes
Completed | 0; 0 eyes | 0; 0 eyes
Not Completed | 327; 327 eyes | 327; 302 eyes

BASELINE CHARACTERISTICS:
Population: Enrolled patients who underwent surgery with an investigational lens in at least one eye.
Units Other Than Participants: Eyes
Groups:
- EVO ICL: Enrolled patients who underwent surgery with an investigational lens in at least one eye
Arm/Group | EVO ICL
Number analyzed (Participants) | 327
Number analyzed (Eyes) | 629
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 327
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213
  Male | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34
  Not Hispanic or Latino | 293
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 11
  White | 274
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 327
Preoperative Manifest Refraction Spherical Equivalent [Mean (Standard Deviation); unit: Diopters] — Mean preoperative Manifest Refraction Spherical Equivalent. Population: 327 participants were enrolled with analysis presented for primary eye (n=327) and fellow eye (n=302)
  Diopters
    Primary Eyes: number analyzed (Eyes) | 327
    Primary Eyes | -7.63 (2.80)
    Fellow Eyes: number analyzed (Eyes) | 302
    Fellow Eyes | -7.61 (2.72)

OUTCOME MEASURES:

1. Primary Outcome: Number of Primary Eyes Requiring Peripheral Iridotomy (PI)
Description: Incidence of PI required to treat elevated intraocular pressure (IOP) caused by mechanical pupillary block in primary eyes.
Time Frame: 6 Months
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Primary Eyes
Number analyzed (Participants) | 327
Number analyzed (Eyes) | 327
eyes | 0

2. Primary Outcome: Endothelial Cell Density (ECD) Change in Primary Eyes.
Description: Endothelial Cell Density (ECD) was determined by analysis of images captured by a specular microscopy device. These images were analyzed by a reading center to determine ECD values before surgery and 6 months after surgery to calculate the mean change (% decrease) of ECD from baseline at month 6 in primary eyes. Negative outcome values represent a reduction in Endothelial Cell Density.
Time Frame: 6 Months
Population: Analysis is based on examination data available at both the pre-operative visit and at the 6-month visit.
Measure: Mean (95% Confidence Interval); unit: percentage change
Units Other Than Participants: Eyes
Arm/Group | Primary Eyes
Number analyzed (Participants) | 321
Number analyzed (Eyes) | 321
percentage change | -2.4 [-2.86 to -1.92]

3. Primary Outcome: Endothelial Cell Density (ECD) <1000 Cells/mm² in Primary Eyes.
Description: Number of eyes with ECD <1000 cells/mm² at month 6 in primary eyes.
Time Frame: 6 months
Population: Analysis is based on examination data available at both the pre-operative visit and at the 6-month visit.
Measure: Number (95% Confidence Interval); unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Primary Eyes
Number analyzed (Participants) | 321
Number analyzed (Eyes) | 321
eyes | 0 [0.00 to 1.14]

4. Primary Outcome: Endothelial Cell Density (ECD) <1500 Cells/mm² in Primary Eyes.
Description: Number of eyes with ECD <1500 cells/mm² at month 6 in primary eyes.
Time Frame: 6 months
Population: Analysis is based on examination data available at both the pre-operative visit and at the 6-month visit.
Measure: Number (95% Confidence Interval); unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Primary Eyes
Number analyzed (Participants) | 321
Number analyzed (Eyes) | 321
eyes | 0 [0.00 to 1.14]

5. Primary Outcome: Number of Ocular Adverse Events (AEs) in Primary Eyes.
Time Frame: 6 Months
Measure: Number; unit: events
Units Other Than Participants: Eyes
Arm/Group | Primary Eyes
Number analyzed (Participants) | 327
Number analyzed (Eyes) | 327
events | 108

6. Secondary Outcome: Number of Primary and Fellow Eyes Requiring Peripheral Iridotomy (PI)
Description: Incidence of PI required to treat elevated intraocular pressure (IOP) caused by mechanical pupillary block in primary and fellow eyes.
Time Frame: 6 Months
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Groups:
- Primary and Fellow Eyes: Primary and fellow implanted eyes
  EVO/EVO+ Visian ICL: The investigational lenses are intended to be implanted within the posterior chamber, directly behind the iris, and in front of the anterior capsule of the human crystalline lens.
Arm/Group | Primary and Fellow Eyes
Number analyzed (Participants) | 327
Number analyzed (Eyes) | 629
eyes | 0

7. Secondary Outcome: Endothelial Cell Density (ECD) Change in Primary and Fellow Eyes.
Description: Endothelial Cell Density (ECD) was determined by analysis of images captured by a specular microscopy device. These images were analyzed by a reading center to determine ECD values before surgery and 6 months after surgery to calculate the mean change (% decrease) of ECD from baseline at month 6 in primary eyes and fellow eyes. Negative outcome values represent a reduction in Endothelial Cell Density.
Time Frame: 6 Months
Population: Analysis is based on examination data available at both the pre-operative visit and at the 6-month visit.
Measure: Mean (95% Confidence Interval); unit: percentage change
Units Other Than Participants: Eyes
Arm/Group | Primary and Fellow Eyes
Number analyzed (Participants) | 321
Number analyzed (Eyes) | 619
percentage change | -2.26 [-2.57 to -1.94]

8. Secondary Outcome: Endothelial Cell Density (ECD) <1000 Cell/mm² in Primary and Fellow Eyes.
Description: Number of eyes with ECD <1000 cell/mm² at month 6 in primary and fellow eyes.
Time Frame: 6 months
Population: Analysis is based on examination data available at both the pre-operative visit and at the 6-month visit.
Measure: Number (95% Confidence Interval); unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Primary and Fellow Eyes
Number analyzed (Participants) | 321
Number analyzed (Eyes) | 619
Eyes | 0 [0.00 to 0.59]

9. Secondary Outcome: Endothelial Cell Density (ECD) <1500 Cell/mm² in Primary and Fellow Eyes.
Description: Number of eyes with ECD <1500 cell/mm² at month 6 in primary and fellow eyes.
Time Frame: 6 months
Population: Analysis is based on examination data available at both the pre-operative visit and at the 6-month visit.
Measure: Number (95% Confidence Interval); unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Primary and Fellow Eyes
Number analyzed (Participants) | 321
Number analyzed (Eyes) | 619
eyes | 0 [0.00 to 0.59]

10. Secondary Outcome: Number of Ocular Adverse Events (AEs) in Primary and Fellow Eyes
Time Frame: 6 Months
Measure: Number; unit: events
Units Other Than Participants: Eyes
Arm/Group | Primary and Fellow Eyes
Number analyzed (Participants) | 327
Number analyzed (Eyes) | 629
events | 203

ADVERSE EVENTS:
Time Frame: 6 months.
Description: Serious Adverse events (SAEs) (ocular and non-ocular) were collected. Non-serious non-ocular adverse events were not collected. The study protocol required that all secondary surgical interventions (SSIs) performed to treat an ocular SAE also be reported as SAEs.
Groups:
- Non-Ocular Serious Adverse Events: Participants who experienced a non-ocular Serious Adverse Event.
Arm/Group | Primary Eyes | Fellow Eyes | Non-Ocular Serious Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/327 | 0/302 | 0/327
Serious Adverse Events (participants affected / at risk) | 10/327 | 6/302 | 2/327
Other Adverse Events (participants affected / at risk) | 82/327 | 65/302 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Eyes (N=327) | Fellow Eyes (N=302) | Non-Ocular Serious Adverse Events (N=327)
Glare/Halo (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Narrow anterior chamber angle (Eye disorders) | 2 (3) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Intraocular lens exchange (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Intraocular lens removal (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Intraocular lens repositioning (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Retinal Surgery (Eye disorders) | 1 (2) | 2 (5) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral Infarction (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Eyes (N=327) | Fellow Eyes (N=302) | Non-Ocular Serious Adverse Events (N=0)
Intraocular pressure increased (Eye disorders) | 75 (77) | 61 (66) | 0 (0)
Anterior chamber cell/flare (Eye disorders) | 7 (7) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated from the study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee are completed. The results of the study may be published or presented by the Investigator(s) after review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed. Prior to publication or presentation, a copy of the final text should be forwarded to Sponsor or designee for comment.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04283149/Prot_SAP_000.pdf